CLINICAL TRIAL: NCT03778060
Title: Cala TWO Device: Clinical Efficacy and Effects on Regional Brain Metabolism in Essential Tremor Subjects Scheduled to Undergo Deep Brain Stimulation Surgery
Brief Title: Long-Term Transcutaneous Stimulation and Essential Tremor: A PET Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Cala Health, Inc. (Industry)
Responsible Party: Principal Investigator, Kendall H. Lee, Clinical Professor, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-006984
Record Dates: First submitted 2018-12-07; First posted 2018-12-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Essential Tremor
Keywords: Transcutaneous Nerve Stimulation; Positron-Emission Tomography
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Masking Description: No other parties will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Transcutaneous stimulation (Experimental): Participants in the clinical study will consist of subjects with essential tremor who are scheduled more than 3 months in advance to undergo deep brain stimulation surgery for treatment of essential tremor at Mayo Clinic. Subjects will wear a Cala TWO stimulator to reduce hand tremors.
  Interventions: Device: Cala TWO stimulator

INTERVENTIONS:
Device: Cala TWO stimulator — Treatment intervention will consist of subjects undergoing 40 minute sessions of transcutaneous stimulation with the Cala TWO stimulator twice daily for 3 months to reduce hand tremors prior to their undergoing deep brain stimulation 'surgery for treatment of essential tremor at Mayo Clinic.

SUMMARY:
Essential tremor (ET) is the most common movement disorder in the United States and affects up to 5% of the population. ET patients experience involuntary shaking of the hands, head and/or voice that can range from mildly limiting to severely disabling.

Treatment options are limited and there are currently no medications specifically designed to treat it, and medications that are prescribed to relieve tremors are often limited by either inadequate efficacy or intolerable side effects. A subset of essential tremor patients whose tremors are inadequately treated by medication choose to undergo deep brain stimulation (DBS) of the ventral intermediate thalamic nucleus. DBS has been shown to be highly effective for tremor suppression. However, DBS carries significant risks. As a result, a very small (less than 3%) percentage of essential tremor patients undergo DBS therapy.

The medical technology company Cala Health has developed a wristband device (the Cala TWO) that offers individuals with essential tremor a novel non-pharmacological, non-invasive alternative, in the form of stimulation of peripheral nerves, to aid in hand tremor relief. This innovative form of therapy has the potential to have important health, quality of life, and economic benefits for essential tremor patients.

The present pilot study (Aim 1) will assess the effectiveness of 3-month twice daily treatment with the Cala TWO device to aid in the relief of hand tremors in adult essential tremor subjects that have been approved to undergo deep brain stimulation surgery at Mayo Clinic - Rochester. This study is a prospective, within subject, non-significant risk study at Mayo Clinic - Rochester, enrolling approximately 20 subjects.

A completely optional component of this study (Aim 2) is seeking to perform three standard PET/CT sessions on a subset of these subjects (n=10) at Mayo Clinic - Rochester to evaluate changes in brain metabolic activity as a result of 3 months treatment with the device. The first session would take place upon a subjects entry into the study (start of month 1) and prior to any treatment with the Cala device, a second the following day after a 40 minute treatment period with the Cala device, and a third session at the end of the third month. This study is a prospective, within subject, greater than minimum risk study.

DETAILED DESCRIPTION:
Hypothesis:

The primary research question is whether customized patterned transcutaneous afferent electrical stimulation to the median and radial nerves via the Cala TWO wrist-band device significantly reduces hand tremors in individuals diagnosed with essential tremor that have been approved as candidates for deep brain stimulation (DBS) surgery. A second research question is whether three months of treatment with the Cala TWO device leads to significant changes in regional brain metabolism that is associated with therapeutic efficacy.

Aims, purpose, or objectives:

Aim 1: Determine the clinical efficacy of the Cala TWO device to transiently reduce hand tremors in the treated hand of subjects with essential tremor (n=20) over a three month treatment period prior to their undergoing DBS surgery for treatment of essential tremor at Mayo Clinic.

Aim 2: Compare regional brain metabolism between baseline, after acute stimulation with the Cala TWO device, and at exit 3 months after therapeutic treatment with the Cala TWO device. 18Ffluorodeoxyglucose (FDG) Positron Emission Tomography (PET)/Computerized Tomography (CT) scans will be applied in a subset (n=10) of essential tremor subjects to evaluate changes in brain tissue metabolic activity corresponding to regional glucose uptake.

Aim 1 Methods:

Design of the Cala TWO device Study: Subjects will be recruited exclusively from adult essential tremor (ET) patients that have been approved by Mayo Clinic Deep Brain Stimulation Group (comprised of neurosurgeons, neurologists, psychiatrists, and radiologists) to undergo deep brain stimulation surgery at Mayo Clinic - Rochester for the treatment of ET. As such, subjects that consent to this study are expected to readily meet the pre-specified inclusion criteria noted below for participation in the study.

Regardless, all subjects will be pre-screened against the inclusion/exclusion criteria through face-to-face interviews. Additionally, baseline function and tremor severity will be collected in the first visit phase of the study. Subjects already taking medications for ET will be permitted these medications during the study with no changes in medication type or dosage.

All subjects will be fitted with a Cala TWO device based on the subject's wrist circumference (small, medium, or large) and stimulation hand (right or left) at the beginning of the study visit. The stimulation hand will be the hand with more severe tremor (or the dominant hand if both hands had equal tremor severity) as determined by the TETRAS task completed during the baseline evaluation and pre-surgery clinical evaluation by the Mayo Clinic DBS group. Once the Cala TWO device has been fitted to the subject's hand a frequency calibration procedure will be conducted in which the subject's tremor frequency will be determined while the subject performs a forward postural hold task. This frequency will then be incorporated into the therapeutic stimulation waveform.

Stimulation will consist of a series of charge balanced biphasic pulses delivered at a frequency of 150 Hz, 300 µs pulse width, and 50 µs inter-pulse period. The stimulation will be alternated between the median and radial nerve at a frequency equal to tremor frequency (i.e. for a measured 5 Hz tremor frequency, stimulation will be applied over the median nerve for 200 msec, then alternated to be applied over the radial nerve for 200 msec). To determine the stimulation amplitude, the site study neurologist will increase the stimulation level by 0.25 mA steps until the subject reports sensation of the stimulus in areas in the hand or finger area. Final stimulation amplitude will be chosen to be the highest level of stimulation below muscle contraction that the subject finds comfortable (mean: 5.4 mA +/- 2.9). Once the maximum tolerable stimulation level has been identified, subjects will receive stimulation at that level during the 40-minute stimulation session. Adverse events will be collected before, during, and after each stimulation session. Subjects will then receive device training and instructions by on-site study personnel for conducting daily home stimulation sessions.

Power Statement: This is a pilot study with a unique subject cohort.

Data Analysis Plan:

An analysis of covariance (ANCOVA) model will be used to assess the statistical significance of the difference in the mean change in tremor before and after treatment.

Efficacy will be measured as the change in the TETRAS scale measure of upper limb tremor following stimulation compared with pre-stimulation. Additional analyses will include the Bain & Findley 4-point scale assessment of typical Activities of Daily Living (ADL) and the Patient Global Impression - Severity (PGI-S) 7-point scale of the subjects' personal assessment of how much their tremor level improved or worsened relative to their baseline state prior to the stimulation session.

The primary safety endpoint will be an analysis of adverse events types and rates for all enrolled subjects, where the adverse event rate will be calculated as the percentage of total subjects with an adverse event.

Aim 2 Methods:

The investigators propose to recruit subjects (n=10; age 21-70) from the population of subjects that have enrolled in the Cala TWO device which is a 3-month treatment duration study with the Cala TWO device prior to subject's scheduled deep brain stimulation surgery. This optional component of this study will perform three standard PET/CT sessions on these subjects at the Mayo Clinic Molecular Research Imaging Facility to evaluate changes in brain tissue metabolic activity as a result of 3 months treatment with the device. The advanced clinical PET scanner PET/CT will be used in this study, equipped with digital silicon photomultiplier detectors.

First session: Takes place upon a subject's entry into the Cala TWO study (start of month 1) and prior to any treatment with the Cala device.

Second session: Takes place the following day after a 40 minute treatment period with the Cala device.

Third session: Takes place at the end of the third month of use of the device.

Minimizing the Radiation Risk: By using an advanced clinical PET scanner, equipped with digital silicon photomultiplier detectors, the investigators will be using a reduced intravenous delivered dose of FDG (8 mCi).

Attenuation Correction Scans: For PET/CT, a low-dose CT fusion skull scan (~1min) will be acquired for attenuation correction and anatomical co-registration.

Step-by-Step Schedule:

The FDG scan slots are available at 7:30am, 8:00am, 8:30am, and 10:30am. Participants with head tremor would present problems in obtaining quality scans. If this is the case, a head secure procedure will be included.

1. A 4 hour fast is required prior to FDG injection. Patients are given instructions to remain well-hydrated and have a low carbohydrate diet 18 hours before their appointment.
2. No significant alcohol or caffeine consumption and no usage of the Cala TWO device within 8 hours of a PET session.
3. Blood sugar level will be checked by a finger-poke blood test. Fasting blood glucose should be under 200 mg/dL.
4. Women of child-bearing potential will go through a urine-pregnancy test, unless there is proof of negative results within 48 hours before the exam.
5. 8 mCi FDG injection through IV and rest at the uptake room (eyes open in a dimly lit room).
6. At 30 minute uptake time, conduct a PET/CT scan for a 15 min. A 1 min CT fusion skull image will be acquired for attenuation correction and anatomical co-registration.

Power Statement: This is a pilot study with a unique subject cohort.

Data Analysis Plan:

CortexID (GE Medical Systems, LLC) and MIMneuro (MIM Software Inc.) will be used to confirm quality control of the PET image. Additional quantitative analysis of PET images will be conducted using SPM, FSL, and Analyze. CortexID. This quantification procedure uses a patient-specific FDG z-score map derived by comparing the surface projection map (z-SPM) with an age- and sex-matched normal control FDG database.

ELIGIBILITY:
Subject population (children, adults, groups): Adults approved for DBS surgery at Mayo Clinic for treatment of essential tremor

Inclusion Criteria:

* Prospective subjects must meet all of the following criteria to be eligible for study participation:
* Must be greater than or equal to 21 years of age. Must be approved for DBS surgery at Mayo Clinic for treatment of essential tremor.
* Competent and willing to provide signed, informed consent to participate in the study.
* Stable dose of tremor medications, if applicable, for 30 days prior to study entry.
* Stable dose of antidepressant medications, if applicable, for 90 days prior to study entry.
* Willing to comply with study protocol requirements including: remaining on a stable dosage of tremor and antidepressant medications, if applicable, during the duration of the study; no significant alcohol or caffeine consumption within 8 hours of study visits; no usage of the Cala TWO device within 8 hours of study visits.

Exclusion Criteria:

* Prospective subjects that meet any of the following criteria are not eligible for enrollment in this study:
* Moderate to severe ethanol dependence as defined by the criteria outlined in the DSM-5 (score of 4 or higher).
* Implanted electrical medical device, such as a pacemaker, defibrillator, or deep brain stimulator.
* Previous thalamotomy procedure, including stereotactic thalamotomy, gamma knife radiosurgical thalamotomy, and focused ultrasound for the treatment of tremor.
* Suspected or diagnosed epilepsy or other seizure disorder. Swollen, infected, inflamed areas, or skin eruptions, open wounds, or cancerous lesions of skin at stimulation site (wrist).
* Peripheral neuropathy affecting the tested upper extremity. Presence of any other neurodegenerative disease like Parkinson plus syndromes suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer's disease.
* Anyone suspected to have the diagnosis of idiopathic Parkinson's disease (PD). This includes excluding anyone with the presence of parkinsonian features including bradykinesia rigidity, or postural instability. Subjects that exhibit only mild resting tremor but no other symptoms or signs of PD may be included.
* Botulinum toxin injection for hand tremor within 6 months prior to study enrollment.
* Are participating or have participated in another interventional clinical trial in the last 30 days which may confound the results of this study, unless approved by the Principal Investigator.
* Significant alcohol or caffeine consumption within 8 hours of study enrollment, which may confound the results of the study, where significant caffeine is considered more than 95 mg (equivalent to a cup of coffee), and significant alcohol is considered more than 14 g (equivalent to 5 oz of wine, 12 oz of beer, or 1.5 oz of distilled spirits).
* Subjects unable to communicate with the investigator and staff. Any health condition that in the investigator's opinion should preclude participation in this study.
* Pregnancy or anticipated pregnancy during the course of the study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Essential Tremor Assessment Following Transcutaneous Stimulation | Patient assessed at entry to study and at exit of study (3 months).
  • The Essential Tremor Rating Assessment Scale (TETRAS) - dominant hand subset mean change (pre-stimulation rating - post-stimulation rating) across visits. Upper limb tremor will be assessed during three maneuvers: forward horizontal reach posture, lateral "wing beating" posture and finger-nose-finger testing. Each upper limb will be assessed and scored individually according to the following scale: 0 = no tremor ; 1 = tremor is barely visible ; 1.5 = tremor is visible, but less than 1 cm ; 2 = tremor is 1- less than 3 cm amplitude ; 2.5 = tremor is 3- less than 5 cm amplitude ; 3 = tremor is 5- less than 10 cm amplitude ; 3.5 = tremor is 10- less than 20 cm amplitude ; 4 = tremor is less than 20 cm amplitude
Assessment of Daily Activities Following Transcutaneous Stimulation | Patient assessed at entry to study and at exit of study (3 months).
  • Bain & Findley Activities of Daily Living (ADL) Scale (pre-stimulation rating - poststimulation rating) across visits. ADL tasks are: Use a spoon to drink soup ; Hold a cup of tea ; Pour milk from a bottle or carton ; Dial a telephone ; Pick up your change in a shop ; Insert an electric plug into a socket ; Unlock your front door with a key. Each task will be rated on a 4-point scale (1-4): 1 = Able to do the activity without difficulty ; 2 = Able to do the activity with a little effort ; 3 = Able to do the activity with a lot of effort ; 4 = Cannot do the activity by yourself
Assessment of Tremor Severity Following Transcutaneous Stimulation | Patient assessed at entry to study and at exit of study (3 months).
  • The Patient Global Impression - Severity scale (PGI-S) on tremor mean improvement change across pre- and post-stimulation sessions. The PGI-S will be a 7-point scale that the participant will use to assess their overall tremor severity of the stimulated hand and consists of: 1 = Normal ; 2 = Hardly perceptible ; 3 = Mild ; 4 = Moderate ; 5 = Marked ; 6 = Severe ; 7 = Extreme

SECONDARY OUTCOMES:
Daily Changes in Tremor over 3 Months of Transcutaneous Stimulation | Patient assessed at entry to study, twice daily over the course of 3 months, and at exit of study (3 months).
  • Kinematic data mean change in units of meters^2/sec (pre-stimulation tremor power - post-stimulation tremor power) across stimulation sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Kendall H Lee, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials